CLINICAL TRIAL: NCT03548506
Title: Subthalamic Steering for Therapy Optimization in Parkinson's Disease
Acronym: SANTOP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital Tuebingen (Other)
Collaborators: Abbott (Industry)
Responsible Party: Principal Investigator, Prof. Dr. Alireza Gharabaghi, Professor, University Hospital Tuebingen
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: SANTOP
Record Dates: First submitted 2018-04-18; First posted 2018-06-07 (Actual); Last update posted 2021-09-29 (Actual); Status verified 2021-09

CONDITIONS: Parkinson Disease
Keywords: STN; DBS; steering; segmented electrode leads
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- STN_O (Active Comparator): Omnidirectional Deep Brain Stimulation of STN
  Interventions: Device: Omnidirectional Deep Brain Stimulation of STN
- STN_D (Experimental): Directional Deep Brain Stimulation of STN
  Interventions: Device: Directional Deep Brain Stimulation of STN

INTERVENTIONS:
Device: Omnidirectional Deep Brain Stimulation of STN — Deep Brain Stimulation
  Arms: STN_O
Device: Directional Deep Brain Stimulation of STN — Deep Brain Stimulation
  Arms: STN_D

SUMMARY:
Twenty patients with idiopathic Parkinson's disease (PD) will be included into this single center randomized controlled double-blind clinical trial (RCT) in a cross-over design. The treatment consists of two different stimulation settings using (i) conventional omnidirectional stimulation of the subthalamic nucleus [STN_O] as active comparator and (ii) directional steering of STN stimulation via a segmented electrode contact [STN_D].

DETAILED DESCRIPTION:
Twenty PD patients will be enrolled in this cross-over double-blind RCT to evaluate both the safety and efficacy of directional STN stimulation [STN_D] compared with standard omnidirectional STN stimulation [STN_O]. The primary outcome measure is objectively quantified muscle rigidity of the upper extremity, i.e., surface EMG recordings of the biceps and triceps muscle during standardized extension/flexion of the elbow joint (Levin et al., 2009) assessed 6 months after implantation in cross-over design. The trial is designed to detect with an 80% power a change of 0.27 mA of the therapeutic stimulation threshold with two-tailed P < 0.05 (Wilcoxon rank sum test). Secondary outcome measures address clinical motor, non-motor, neurocognitive and neuropsychiatric symptoms, freezing of gait, and quality of life. Visits are scheduled at weeks 1 (V1), 6 (V2), 24 (V3), 27 (V4), and 30 (V5) from baseline (V0).

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Idiopathic Parkinson's disease (according to the "British Brain Bank criteria" (Hughes, 1992) including genetic forms

Exclusion Criteria:

* Cognitive impairment (Mini Mental State Exam < 20)
* Suicidality, Psychosis
* Other severe pathological chronic condition that might confound treatment effects or interpretation of the data
* Pregnancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-04-19 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2022-04 (Estimated)

PRIMARY OUTCOMES:
Muscle Rigidity | 6 months post-operatively
  Surface-Electromyography (EMG) of M. biceps brachii and M. triceps brachii

SECONDARY OUTCOMES:
Clinical motor and non-motor symptoms (1) | 6 months post-operatively
  MDS-UPDRS I
Clinical motor and non-motor symptoms (2) | 6 months post-operatively
  MDS-UPDRS II
Clinical motor and non-motor symptoms (3) | 6 months post-operatively
  MDS-UPDRS III
Clinical motor and non-motor symptoms (4) | 6 months post-operatively
  MDS-UPDRS IV
Clinical motor and non-motor symptoms (5) | 6 months post-operatively
  Bradykinesia evaluation
Clinical motor and non-motor symptoms (6) | 6 months post-operatively
  Tremor evaluation
Clinical motor and non-motor symptoms (7) | 6 months post-operatively
  Deep brain stimulation impairment scale (DBS-IS):
  * the scale consists of 22 questions and 6 subscales;
  * subscales: 1. postural instability and gait difficulties (range 0-20), 2. cognitive impaiment (range 0-20), 3. speaking problems (range 0-12), 4. apathy (range 0-12), 5. impulsivity (range 0-12), and 6. difficulties related to DBS device (range 0-12);
  * Ʃ 1-6 DBS-IS total range: 0-88;
  * Ʃ 1-5 DBS-IS total range: 0-76;
  * higher values represent worsening of symptoms
Clinical motor and non-motor symptoms (8) | 6 months post-operatively
  Clinical global impression self
Neurocognitive and non-motor symptoms (1) | 6 months post-operatively
  Modulation range
Neurocognitive and non-motor symptoms (2) | 6 months post-operatively
  Spatial with a visual Odd-Ball test
Neurocognitive and non-motor symptoms (3) | 6 months post-operatively
  Verbal Working Memory with an auditory Odd-Ball test
Neurocognitive and non-motor symptoms (4) | 6 months post-operatively
  Power of Attention (Cognitive Drug Research Battery)
Neurocognitive and non-motor symptoms (5) | 6 months post-operatively
  Digit Vigilance Accuracy (Cognitive Drug Research Battery)
Neurocognitive and non-motor symptoms (6) | 6 months post-operatively
  Executive functions with One Touch Tower of London (Cambridge Neuropsychological Test Automated Battery, CANTAB)
Neurocognitive and non-motor symptoms (7) | 6 months post-operatively
  Montreal Cognitive Assessment (MoCA)
Neuropsychiatric symptoms (1) | 6 months post-operatively
  Beck Depression Inventory (BDI)
Neuropsychiatric symptoms (2) | 6 months post-operatively
  Apathy Scale/Lille Apathy rating scale/Neuropsychiatric inventory
Freezing of gait (1) | 6 months post-operatively
  Capsit-PD
Freezing of gait (2) | 6 months post-operatively
  Freezing of Gait Assessment Course
Quality of life | 6 months post-operatively
  Parkinson's Disease Questionaire (PDQ-39)

OTHER OUTCOMES:
Electroencephalography | up to 6 months post-operatively
  Electroencephalography (EEG)
Electromyography | up to 6 months post-operatively
  Electromyography (EMG)

CONTACTS AND LOCATIONS:
Overall Officials: Alireza Gharabaghi, MD, Principal Investigator — Division of Functional and Restorative Neurosurgery, Department of Neurosurgery, Tuebingen, Germany; Daniel Weiss, MD, Principal Investigator — Department for Neurodegenerative Diseases, Centre for Neurology, Tuebingen, Germany, and Hertie-Institute for Clinical Brain Research
Locations (1):
- University Hospital Tuebingen, Dep. of Neurosurgery (Functional Neurosurgery) and Neurology (Neurodegenerative Diseases), Tübingen, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Levin J, Krafczyk S, Valkovic P, Eggert T, Claassen J, Botzel K. Objective measurement of muscle rigidity in Parkinsonian patients treated with subthalamic stimulation. Mov Disord. 2009 Jan 15;24(1):57-63. doi: 10.1002/mds.22291. PMID 18855925
- [Derived] Gharabaghi A, Cebi I, Leavitt D, Scherer M, Bookjans P, Brunnett B, Milosevic L, Weiss D. Randomized crossover trial on motor and non-motor outcome of directional deep brain stimulation in Parkinson's disease. NPJ Parkinsons Dis. 2024 Oct 26;10(1):204. doi: 10.1038/s41531-024-00812-0. PMID 39461964